CLINICAL TRIAL: NCT05636774
Title: Empower the Heart of Patients With Terminal Cancer Using Cardiac Medicines Trial - EMPATICC (INCOR1)
Brief Title: Empower the Heart of Patients With Terminal Cancer Using Cardiac Medicines Trial
Acronym: EMPATICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Charite University, Berlin, Germany (Other); Universitätsklinikum Leipzig (Other); University Hospital Heidelberg (Other); University Hospital Homburg/Saar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-10545-AF
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Patients With Advanced Cancer Receiving Specialized Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Note: We involve blinded and unblinded study investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart failure medication arm (Experimental): Combination of Sacubitril/valsartan, Ivabradine, Ferric carboxymaltose and/or Empagliflozin
  Interventions: Drug: Heart failure medication
- Placebo arm (Placebo Comparator): Placebo tables / infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Heart failure medication — Combination of Sacubitril/valsartan, Ivabradine, Ferric carboxymaltose and/or Empagliflozin.
  Arms: Heart failure medication arm
Drug: Placebo — Placebo tables / infusion
  Arms: Placebo arm

SUMMARY:
The pathophysiological implications of various cancer diseases and anti-cancer therapies is the occurrence of a cardiac disease-like phenotype with cardiac dysfunction, cardiac wasting, and cardiac homeostasis changes (incl. fibrosis and apoptosis) in end-stage cancer patients, causing heart failure like syndrome with development of congestion, dyspnoea and severely reduced physical functioning. The present trial aims to evaluate, if a heart failure medication improves the self-care ability and self-reported health care status of patients with with advanced cancer receiving specialized palliative care.

ELIGIBILITY:
Inclusion criteria:

Basic Criteria:

* Patients with solid cancer in Union internationale contre le cancer (UICC) stage 4 (in palliative care)
* 1-6 months expected survival as assessed according to local standards
* Patients under optimised analgetic therapy

Group 1 Criteria:

* Heart rate >70 bpm
* NT-proBNP >600 pg/ml
* Elevated high-sensitive troponin (>99th percentile of respective test)
* LVEF <55%
* Heart failure with preserved ejection fraction (HFpEF) likelihood medium or large
* Evidence of left ventricular (LV) mass reduction >15% since start of cancer
* Iron deficiency (ID) with transferrin saturation (TSAT) <20%

Group 2 Criteria:

* 4 m walking time (>=6.0 secs for 4m - test will be performed twice and the average time is calculated) or not able to walk 4m at all.
* Not being able to wash oneself in at least 3 of the last 7 days
* Presence of shortness of breath (SoB) (NYHA IV)

Requirement for inclusion:

At least two fulfilled criteria of Group 1 PLUS at least one fulfilled criterion of Group 2

Exclusion criteria:

* Previous participation in this trial. Participation is defined as randomised
* Ongoing haemodialysis
* Patients currently on intravenous iron
* Acute sepsis with at least 2 points at the quick sequential organ failure assessment (qSOFA) score. The use of i.v.-antibiotics is permitted in patients with a lower qSOFA score.
* Ongoing acute exacerbation of chronic obstructive pulmonary disease (COPD) Acute ST elevation myocardial infarction (STEMI) or severe pulmonary embolism (PE) or severe deep vein thrombosis (DVT) (currently or in last 4 weeks)
* Current uncontrolled cerebral metastasis
* Impaired neurological status, precluding the ability to walk
* Unable or unwilling to give written informed consent
* Participation in other interventional trials using investigational products in randomised settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Win ratio with the following 3 hierarchical components: (1) days alive and able to wash oneself, (2) ability to walk 4m, (3) self-reported patient global assessment of subjective well-being, during the 30-day placebo-controlled phase | since baseline during 30 days of follow-up
  The primary endpoint is analyzed using the win ratio approach, comparing patient pairs based on the hierarchy of the following 3 components:
  1. The first component, "days alive and able to wash themselves," was assessed over a 30 ± 2-day period, with counts ranging from 0 to 32 days.
  2. The second component, "ability to walk 4 meters," was assessed at Days 10, 20, and 30, with counts ranging from 0 to 3 visits.
  3. The third component, "self-reported PGA of subjective well-being," was assessed at the last common assessment visit where both patients were alive (Day 30, 20, or 10) using a 7-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No